CLINICAL TRIAL: NCT04375241
Title: Detection of Asymptomatic Atrial Fibrillation in Persons of 65 Year of Age or Older
Acronym: DETECT AF
Status: Completed | Type: Observational
Sponsor: Diagram B.V. (Other)
Responsible Party: Sponsor
Other Study IDs: 9275
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: Mobile ECG device; Asymptomatic atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening with Mobile ECG Device: Subjects with asymptomatic atrial fibrillation will be screened by using a Mobile ECG Device
  Interventions: Other: Subjects with asymptomatic atrial fibrillation will be screened by using a Mobile ECG Device

INTERVENTIONS:
Other: Subjects with asymptomatic atrial fibrillation will be screened by using a Mobile ECG Device — Subjects with asymptomatic atrial fibrillation will be screened by using a Mobile ECG Device

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia. Although the condition itself is not life-threatening, the complications result in increased morbidity and mortality. AF is often asymptomatic and a considerable number of people suffering from AF are not aware of their condition. Unfortunately, a cerebral infarction is often the first clinical manifestation. The idea to screen subjects opportunistically for Asymptomatic Atrial Fibrillation (AAF) was infeasible until recently. However, with a recently-developed smartphone connected Mobile ECG Device (MED), this seems to be feasible after all.

The main objectives are:

* To examine the feasibility of screening subjects of ≥65 years old for AAF.
* To validate the smartphone connected MED as an AAF screening instrument for application in transmural care in the Netherlands.

DETAILED DESCRIPTION:
Study design:

Prospective validation study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Is willing to give informed consent

Exclusion Criteria:

* Known medical history with Atrial Fibrillation
* Not mental competent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The participants of this study will be subjects who visit their general practicioner or cardiologist or who visit the DETECT AF team at an event.
Sampling Method: Non-Probability Sample
Enrollment: 2168 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the mobile ECG device | At screening
Specificity of the mobile ECG device | At screening

CONTACTS AND LOCATIONS:
Locations (1):
- Isala, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided to share the individual participant data.